CLINICAL TRIAL: NCT00298584
Title: Comparison of Infant Pain Responses Between Two Different Methods of Urine Collection for Diagnosis of Infection: Suprapubic Aspiration and Urinary Catheterization
Brief Title: Comparison of Infant Pain Responses Between Two Different Methods of Urine Collection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1000008396
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2007-02-23 (Estimated); Status verified 2006-08

CONDITIONS: Pain; Intensive Care, Neonatal
Keywords: Diagnostic techniques, urological; urinary catheterization; Aspiration; Neonates; Neonatal Intensive Care Unit; Infant, Newborn; Infant, Premature; Infant, Low-birth weight
MeSH Terms: conditions — Pain; Premature Birth | interventions — Urinary Catheterization

INTERVENTIONS:
Procedure: Percutaneous Suprapubic Aspiration
Procedure: Urethral Catheterization

SUMMARY:
The purpose of this study is to determine which of the two procedures commonly used to collect urine, percutaneous suprapubic aspiration (SPA) and urethral catheterization (UC), is less painful, and the success rates and complication rates associated with both methods.

DETAILED DESCRIPTION:
Infants hospitalized in the NICU undergo numerous invasive and painful procedures. Exposure to early repeated painful procedures has been correlated with both short-term and long-term negative sequelae, such as altered pain responses and increased sensitivity to pain (Taddio 2005). Fifty eligible infants in the NICU will be randomized to undergo urine collection by either suprapubic aspiration (SPA) or urinary catheterization (UC). Outcome measures will include pain, procedure success, and procedure duration. Pain will be measured using facial grimacing (the infant's face will be videotaped for the entire procedure), heart rate and oxygen saturation. Procedure success will be defined by the collection of about 2mL of urine (Falcao, 1999). The procedure duration in seconds for the first attempt will be calculated. Infants will be monitored during the procedure for adverse events such as apnea, bradycardia, desaturation, emesis, increased ventilatory support. Results will be extremely valuable in aiding health care providers to choose a urine collection technique that minimizes the pain and maximizes the success of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the Neonatal Intensive Care Unit (NICU) who require urine samples for microbiological analysis

Exclusion Criteria:

* Clinical diagnosis of birth asphyxia or seizures
* Neurological conditions
* Congenital anomalies associated with the central nervous system, gut, or genitourinary tract
* Abdominal distension or abdominal infection/cellulitis
* Colostomy
* Inguinal hernia
* Organomegaly
* Bleeding diatheses (thrombocytopenia or coagulopathy)
* Receiving analgesics or sedatives

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2006-02

PRIMARY OUTCOMES:
infant pain response, as measured by facial grimacing and changes in heart rate and oxygen saturation during the procedure

SECONDARY OUTCOMES:
success rate of obtaining a sample suitable for analysis
adverse events, such as post-procedure haematuria, haemorrhage, haematoma, peritonitis, bowel perforation, abdominal wall abscess, and induction of infection, bladder perforation, urethral knots
success rate of procedure according to infant factors; gestational age and sex

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] El-Naggar W, Yiu A, Mohamed A, Shah V, Manley J, McNamara P, Taddio A. Comparison of pain during two methods of urine collection in preterm infants. Pediatrics. 2010 Jun;125(6):1224-9. doi: 10.1542/peds.2009-3284. Epub 2010 May 17. PMID 20478939